CLINICAL TRIAL: NCT01599468
Title: Effects of Tranexamic Acid on Post Partum Hemorrhage by Uterine Atony After Cesarean Section Delivery: a Randomized, Placebo Controlled Trial.
Brief Title: Can Tranexamic Acid Reduce Bleeding After Post Partum Hemorrhage in Cesarean Section Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hédi Chaker Hospital (Other)
Responsible Party: Principal Investigator, mohamed ayedi, Principal Investigator, Hédi Chaker Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TXA-1
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Post Partum Hemorrhage
Keywords: post partum hemorrhage; transfusion; tranexamic acid
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tranexamic acid, post partum hemorrhage (Experimental)
  Interventions: Drug: Tranexamic Acid
- placebo (Placebo Comparator)
  Interventions: Drug: saline serum

INTERVENTIONS:
Drug: Tranexamic Acid — 10 mg/kg of tranexamic acid as induction dose within 12 minutes and 1mg/Kg/h as maintenance within the 2 following hours
  Other Names: exacyl
  Arms: tranexamic acid, post partum hemorrhage
Drug: saline serum — The Placebo group received normal saline with the same volumes
  Other Names: normal saline; NaCl 0.9%
  Arms: placebo

SUMMARY:
The purpose of this study was to evaluate the effect of early administration of tranexamic acid (TXA) on post partum hemorrhage caused by uterine atony after cesarean section delivery.

This was a randomised, placebo controlled trial including 74 patients. The investigators included ASA1 parturients with correct haemostatic status undergoing cesarean section under spinal anesthesia. The randomization begins after the inefficacy of oxytocin injections and starting up sulprostone perfusion at the request of the surgeon. TXA Group received 10 mg/kg of tranexamic acid as induction dose within 12 minutes and 1mg/Kg/h as maintenance within the 2 following hours. Placebo Group received same volumes of normal saline. The investigators compared blood loss and transfusions in both groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA1 parturients
* aged from 20 to 40
* correct preoperative haemostatic status (prothrombine ratio > 60 % and platelet rate > 100 000),
* cesarean section under spinal anesthesia complicated by uterine atony needing the introduction of Sulprostone

Exclusion Criteria:

* abnormal placentation
* severe pre-eclampsia
* coagulopathy and uterine rupture
* the contra indications of TXA : past history of vascular occlusive event, convulsion, and allergy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
volume blood loss | within 5 days after delivery

SECONDARY OUTCOMES:
transfusion rates. | within 5 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: mohamed ayedi, Principal Investigator — hedi chaker university hospital of sfax, tunisia
Locations (1):
- Hedi Chaker University Hospital of Sfax, Department of Anesthesiology and Intensive Care, Sfax, Sfax Governorate, Tunisia

REFERENCES:
- [Background] Ducloy-Bouthors AS, Jude B, Duhamel A, Broisin F, Huissoud C, Keita-Meyer H, Mandelbrot L, Tillouche N, Fontaine S, Le Goueff F, Depret-Mosser S, Vallet B; EXADELI Study Group; Susen S. High-dose tranexamic acid reduces blood loss in postpartum haemorrhage. Crit Care. 2011;15(2):R117. doi: 10.1186/cc10143. Epub 2011 Apr 15. PMID 21496253